CLINICAL TRIAL: NCT04566809
Title: Cognitive Approach Using Functional Electric Stimulation for Grasp and Pinch Rehabilitation in Persons Affected by Cervical Spinal Cord Injury, a Randomized Controlled Trial
Brief Title: Cognitive Rehabilitation and FES for Hand Functionality in Persons With Cervical Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Matteo Olivieri, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 3879A
Record Dates: First submitted 2020-09-14; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injury at C5-C7 Level
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: FES+CBA (Experimental): FES+CBA participants executed FES and CBA treatment which means that during the stimulation they manipulated different tools. In particular, for the first ten sessions the participants were invited to manipulate specific objects: squares, rectangles and pyramids of different sizes; touch on plastic test tubes coated with materials of different consistency; these two exercises were performed both with open and closed eyes. Finally, for the last ten sessions the participants were asked to execute specific tasks, depending on person's life before the lesion.
  Interventions: Other: FES+CBA
- Control Group: FES (Active Comparator): FES participants received only FES to improve their manipulating skills without the interaction with objects, but only with the muscle contraction induced by the devices.
  Interventions: Other: FES

INTERVENTIONS:
Other: FES+CBA — The experimental treatment was formerly composed by 20 sessions of FES for the hand in combination with a structured cognitive therapy
  Other Names: Functional Electric Stimulation, Cognitive Therapy
  Arms: Experimental group: FES+CBA
Other: FES — The control treatment was formerly composed by 20 sessions of FES for the hand
  Other Names: Functional Electric Stimulation
  Arms: Control Group: FES

SUMMARY:
16 persons affected by Cervical-SCI were recruited for the study and randomly assigned to the Control Group (CG) or to the Experimental Group (EG). Persons of the CG (n = 8) executed 20 sessions of FES for the rehabilitation of hand functions (grasp or pinch), participants of the EG (n = 8) performed 20 sessions of FES and CBA in addition. The primary assessment was a modified version of Bimanual Activity Test (10 tasks); also, SCIM-II and measurement of grasping strength only in participants submitted to grasp rehabilitation were evaluated.

DETAILED DESCRIPTION:
Each participant followed twenty sessions of hand rehabilitation, three times per week. Each treatment, for both CG and EG, lasted about forty minutes.

The FES devices chosen for this research stimulated "grasp" or "pinch" function: the NESS H200 (NESS Ltd., Ra'anana, Israel) was used if patient needed to improve the grasp functions, otherwise the Microstim (Microstim, Medel, Hamburg, Germany) was used to increase pinch functions. In order to provide FES, the five electrodes of NESS H200 were first humidified with warm water and then inserted in the right size place of the rigid splint worn by the patient, while Microstim was used with four standard electrodes, two for each muscle treated. In both case the stimulation was triggered by the therapist clicking a button (Table 1).

The participants of CG received only FES to improve their manipulating skills without the interaction with objects, but only with the muscle contraction induced by the devices.

The participants of EG executed FES and CBA treatment which means that during the stimulation they manipulated different tools. In particular, for the first ten sessions the participants were invited to manipulate specific objects: squares, rectangles and pyramids of different sizes; touch on plastic test tubes coated with materials of different consistency; these two exercises were performed both with open and closed eyes. Finally, for the last ten sessions the participants were asked to execute specific tasks, depending on person's life before the lesion.

ELIGIBILITY:
Inclusion Criteria:

* C-SCI with neurological level between C2-T1;
* reduced ability of hand functions;
* excitable muscles and FES tolerability.

Exclusion Criteria:

* any trauma or surgery to the target hand or upper limb within the last 12 months,
* amputation of any digits on the target hand,
* severe spasticity in the target hand or upper limb preventing use of the instruments,
* experienced autonomic dysreflexia or hypotension in response to FES,
* any contraindication to FES such as: cardiac pacemaker, epilepsy, forearm fracture, pregnancy, skin lesions, cancer or tumor, intracranial metal implants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-21 (Actual)

PRIMARY OUTCOMES:
Performance test: Bimanual Ability Test (BAT) | 2 years
  10 items evaluated, each one from 0 to 60 seconds. Less time needed means better skills

SECONDARY OUTCOMES:
Spinal Cord Independence Measure (SCIM) | 2 years
  The score varies from 0 to 100. Higher the score, patient more independent in its daily life
Grasping Strength (GS) | 2 years
  Grasping Strength evaluated with a dynamometer (from 1 to 90 kg) more kg means more strength

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP